CLINICAL TRIAL: NCT03654040
Title: A Phase I/II Drug Withdrawal Study of Alloantigen-Specific Tregs in Liver Transplantation
Brief Title: Liver Transplantation With Tregs at UCSF
Acronym: LITTMUS-UCSF
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated by the Sponsor prior to any participants receiving the investigational product.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN074ST; UM1AI109565 (NIH); NIAID CRMS ID#: 38481 (Other: DAIT NIAID)
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Liver Transplant
Keywords: alloantigen-reactive Tregs (arTreg); immunosuppression; operational tolerance
MeSH Terms: interventions — Leukapheresis; Blood Component Removal; Cyclophosphamide; Mesna; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- arTreg (Experimental): arTreg: alloantigen-reactive T regulatory cells
  The investigational product is donor alloantigen-reactive regulatory T cells (arTreg). Supportive regimen for receipt of arTregs includes everolimus, leukapheresis, cyclophosphamide, and mesna.
  Note: Participants who receive at least the minimum Treg product (arTreg) dose of 30 to <90 x10^6 total cells will be included in intent-to-treat analysis.
  Interventions: Biological: arTreg; Procedure: leukapheresis; Drug: cyclophosphamide; Drug: mesna; Drug: everolimus

INTERVENTIONS:
Biological: arTreg — Eligible participants will receive a single dose of Treg product (arTreg). The target dose is at least 90 x 10^6 total cells.
  Method of receipt: peripheral intravenous (IV) infusion, administered over 20 to 30 minutes.
  Other Names: donor alloantigen-reactive regulatory T cells; CD4+CD25+CD127[lo] Treg cells
Procedure: leukapheresis — Leukapheresis will be the method employed to recover peripheral blood mononuclear cells (PBMCs) from the allograft recipient. The recipient will undergo the procedure prior to initiating the cyclophosphamide conditioning regimen.
  Procedure on Day -3 (-1 day) prior to Treg product (arTreg) IV infusion.
  Other Names: apheresis
Drug: cyclophosphamide — 40 mg/kg administered intravenously (IV) following leukapheresis and between 1 to 3 days prior to Treg product (arTreg) infusion, per institutional standard of care.
  Other Names: Cytoxan®; CTX
Drug: mesna — Mesna is administered:
  * Intravenously to inhibit hemorrhagic cystitis induced by cyclophosphamide, and
  * In conjunction with the cyclophosphamide, per institutional practice with CTX.
  Other Names: Mesnex®
Drug: everolimus — EVR is approved for prophylaxis of allograft rejection in adults receiving a liver transplant. Per protocol: Post transplantation, subject will initially receive standard IS with tacrolimus (TAC),plus a mycophenolate product and/or steroids.Subsequently, evaluation for eligibility to be converted to EVR-based IS regimen will occur and, when applicable, proceed. Once the optimal EVR trough level is achieved,TAC dose will be reduced. When target EVR and TAC levels are maintained over two consecutive measurements, ALT liver function test (LFT) is ≤50 U/L, GGT LFT is ≤ the upper limit of normal or ≤ 1.5 times the baseline GGT, subject will be considered successfully converted to EVR-based IS regimen. EVR doses will be administered/monitored/adjusted over time.
  Other Names: EVR; Afinitor®; Zortress®

SUMMARY:
This is a single-center, prospective, open-label, non-randomized clinical trial exploring cellular therapy to facilitate immunosuppression withdrawal in liver transplant recipients.

DETAILED DESCRIPTION:
The researchers in this study plan to enroll 9 participants. Eligible participants will receive a single dose of Treg product (arTreg). The target dose is at least 90 to 500 x 10^6 total cells.

Participants who successfully withdraw from all immunosuppression (IS) will undergo a research biopsy at 52 weeks following IS discontinuation to determine whether they meet the primary efficacy outcome of operational tolerance. Participants determined to be operationally tolerant will be followed until 104 weeks following IS discontinuation. Participants who fail drug withdrawal after 52 weeks but before 104 weeks will be followed until week 104 or 12 weeks after resuming immunosuppression, whichever is longer.

Participants who do not successfully withdraw from all IS will complete 104 weeks of High Intensity Safety Follow-up after failing immunosuppression withdrawal.

*** IMPORTANT NOTICE: *** The National Institute of Allergy and Infectious Diseases and the Immune Tolerance Network do not recommend the discontinuation of immunosuppressive therapy for recipients of cell, organ, or tissue transplants outside of physician-directed, controlled clinical studies. Discontinuation of prescribed immunosuppressive therapy can result in serious health consequences and should only be performed in certain rare circumstances, upon the recommendation and with the guidance of your health care provider.

ELIGIBILITY:
Inclusion Criteria:

Eligibility:

Recipient:

* Individuals must meet all of the following criteria to be eligible for this study:

  1. Able to understand and provide informed consent
  2. End-stage liver disease and listed for a living or deceased-donor primary solitary liver transplant
  3. Agreement to use contraception
  4. For candidates with a history of hepatitis C virus (HCV), completed treatment for HCV, maintaining a sustained viral response of ≥24 weeks duration by the day of transplant
  5. Positive Epstein-Barr virus (EBV) antibody test, and
  6. Immunizations are up-to-date based on the Advisory Committee on Immunization Practices (ACIP) recommendations for individuals with Liver Disease and Adult Vaccination, unless the investigator determines that administering a recommended immunization is not in the patient's best interest.

     Living Donor:
* Living donors must meet all of the following criteria to be eligible for this study:

  1. Able to understand and provide informed consent
  2. Meets site-specific clinical donor eligibility requirements
  3. Meets donor eligibility manufacturing requirements within 7 days before or after the blood collection for manufacturing, and
  4. Willingness to donate appropriate biologic samples.

Deceased Donor:

Deceased donors must meet the following criteria for their recipients to remain eligible:

1. Meets site-specific clinical donor eligibility requirements and
2. Meets donor eligibility manufacturing requirements.

Note:

* There are several stages to this study.
* Eligibility is evaluated at many time points during the study to assess whether a participant is safe to proceed to the next study stage.

Exclusion Criteria:

Recipient:

* Individuals who meet any of the following criteria will not be eligible for this study:

  1. History of previous organ, tissue or cell transplant
  2. For cytomegalovirus (CMV) antibody negative recipients, a (CMV) antibody positive donor
  3. Known contraindication to cyclophosphamide or mesna
  4. Serologic evidence of human immunodeficiency virus (HIV)-1/2 infection
  5. The need for chronic anti-coagulation or anti-platelet agents other than aspirin that cannot be safely discontinued for a minimum of 1 week to safely perform a liver biopsy
  6. End stage liver disease secondary to autoimmune etiology (autoimmune hepatitis, primary biliary cirrhosis, or primary sclerosing cholangitis) or other contraindications to drug withdrawal
  7. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up visit schedule
  8. Any condition that, in the opinion of the investigator, may interfere with study compliance
  9. History of cardiac disease (ischemic heart disease requiring revascularization, history of or current treatment for dysrhythmia, or evidence of congestive heart failure), unless cleared by a cardiologist
  10. Any past or current medical problems, treatments or findings that are not listed above, which, in the opinion of the investigator, may:

      * pose additional risks from participation in the study,
      * interfere with the candidate's ability to comply with study requirements, or
      * impact the quality or interpretation of the data obtained from the study.

        * This includes past, present or future enrollment in studies that affect eligibility at the time of everolimus (EVR) conversion
  11. History of malignancy or any concomitant malignancy, except:

      * hepatocellular carcinoma,
      * completely treated in-situ cervical carcinoma, or
      * completely treated basal cell carcinoma.
  12. Chronic use of systemic glucocorticoids or other immunosuppressives, or biologic immunomodulators.

      Living Donor:
* There are no exclusion criteria for living donors.

Deceased Donor:

-There are no exclusion criteria for deceased donors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Feng, MD, PhD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: The aim is to share data available to the public within 24 months upon completion of the study.
Access Criteria: ImmPort public data access.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network web site — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 prospective transplant recipients and 12 living donors were enrolled from a single study center in the US between April 2021 and February 2023. The study was terminated by the sponsor in February 2023 prior to any participant receiving the investigational product, arTregs.
Pre-assignment Details: Participants were enrolled prior to transplant & had to wait for an available liver which was received per the institution's standard of care. If recipient rec'd a liver from a living donor, the donor also enrolled into the study to collect biological samples to aid in the manufacturing of the investigation product, arTregs. Immunosuppression medication was required to be stabilized and converted from tacrolimus to everolimus prior to transplant recipient receiving the investigational product
Groups:
- Enrolled Transplant Recipient, Did Not Receive arTregs: These participants were prospective transplant recipients who were consented and enrolled into the study, but did not receive arTregs.
- Enrolled Living Donor: These participants were living donors of the prospective transplant recipient who consented and enrolled into the study.
Period: Overall Study
Arm/Group | Enrolled Transplant Recipient, Did Not Receive arTregs | Enrolled Living Donor
Started | 30 | 12
Completed | 0 | 5
Not Completed | 30 | 7
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study terminated by sponsor | 8 | 2
Not completed — Failure to initiate study therapy | 2 | 0
Not completed — Transplanted at another center | 2 | 0
Not completed — Failure to meet eligibility criteria | 14 | 2
Not completed — No longer transplant candidate | 1 | 0
Not completed — Manufacturing unable to accept specimens | 1 | 0
Not completed — Recipient ineligible | 0 | 2
Not completed — Received deceased liver | 0 | 1

BASELINE CHARACTERISTICS:
Population: Transplanted participants who enrolled but did not receive arTregs and living donors of the prospective transplant recipient who consented and enrolled into the study
Groups:
- Enrolled, Transplant Recipient Did Not Receive arTregs: These participants were consented and enrolled into the study but did not receive arTregs.
- Total: Total of all reporting groups
Arm/Group | Enrolled, Transplant Recipient Did Not Receive arTregs | Enrolled Living Donor | Total
Number analyzed (Participants) | 30 | 12 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (10.35) | 37.3 (14.09) | 49.9 (13.69)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: <=18 years | 0 | 0 | 0
  Age, Categorical: Between 18 and 65 years | 26 | 11 | 37
  Age, Categorical: >=65 years | 4 | 0 | 4
  Age, Categorical: Missing | 0 | 1 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 18 | 5 | 23
  Unknown | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 24 | 8 | 32
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 9 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 30 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Adverse Events (AEs) Attributed to the Investigational Product, arTreg
Description: * AEs will be attributed to alloantigen-reactive Tregs (arTreg) when the AE is reported with possible or related attribution to arTreg.
  * Grading: According to the NCI Common Terminology Criteria for Adverse Events Manual [NCI-CTCAE version 5.0, published November 27, 2017].
Time Frame: From arTreg infusion through completion of study participation
Population: Data were not collected. The study was terminated prior to any participant receiving the investigational product, arTregs. The study's low enrollment would not allow for study completion within the necessary timeframe.
Groups:
- Enrolled, Received arTregs: These participants were consented and enrolled into the study and received arTregs.
Arm/Group | Enrolled, Received arTregs
Number analyzed (Participants) | 0

2. Primary Outcome: Number and Severity of Adverse Events (AEs) Attributed to Supportive Regimen: Leukapheresis, Cyclophosphamide or Mesna
Description: * AEs will be attributed to the supportive regimen for this study when the AE is reported with possible or related attribution to leukapheresis, cyclophosphamide, or mesna.
  * Grading: According to the NCI Common Terminology Criteria for Adverse Events Manual [NCI-CTCAE version 5.0, published November 27, 2017].
Time Frame: From ≤3 days prior to arTreg infusion through completion of study participation (Up to 3 months)
Population: These participants were consented and enrolled into the study and received at least part of the supportive regimen of leukapheresis, cyclophosphamide, or mesna.
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled, Received Supportive Regimen: These participants were consented and enrolled into the study and received at least part of the supportive regimen of leukapheresis, cyclophosphamide, or mesna.
Arm/Group | Enrolled, Received Supportive Regimen
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: Number of Operationally Tolerant Participants
Description: Operational tolerance is defined as:
  * Discontinuation of all immunosuppression (IS) for 52 weeks,
  * Alanine aminotransferase (ALT) and gamma-glutamyl transpeptidase (GGT) ≤ 50 U/L for ≥ 2 measurements separated by ≥1 week in the 6 weeks prior to the liver biopsy at 52 weeks after the last IS dose, and
  * Liver biopsy at 52 weeks (±4 weeks) after the last IS dose that meets the biopsy criteria for operational tolerance, as assessed by central pathology.
Time Frame: 52 (± 4 weeks) after the last dose of immunosuppression
Population: as for outcome 1
Arm/Group | Enrolled, Received arTregs
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants Who Develop a Malignancy
Description: The number of participants that are diagnosed with malignancy, any type.
Time Frame: Time of enrollment through completion of study participation (Up to 1.8 years)
Population: Participants who enrolled, but did not receive arTregs
Measure: Number; unit: participants
Groups:
- Enrolled, Did Not Receive arTregs: These participants were consented and enrolled into the study but did not receive arTregs.
Arm/Group | Enrolled, Did Not Receive arTregs
Number analyzed (Participants) | 30
participants | 1

5. Secondary Outcome: Incidence of ≥Grade 3 Infections Following arTreg Infusion
Description: Grading: According to the NCI Common Terminology Criteria for Adverse Events Manual [NCI-CTCAE version 5.0, published November 27, 2017].
Time Frame: From arTreg infusion through completion of study participation
Population: as for outcome 1
Arm/Group | Enrolled, Received arTregs
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Biopsy-Proven Acute Rejection (AR) and/or Clinical Rejection Events at Any Time After Alloantigen-Reactive Tregs (arTreg) Infusion
Description: Definitions:
  * AR: Diagnosed in accordance with Banff global assessment criteria
  * Clinical Rejection: Participants who are treated empirically based on investigator clinical suspicion in cases where a biopsy is indeterminate or in rare cases, where a biopsy cannot be performed.
Time Frame: From arTreg infusion through completion of study participation
Population: as for outcome 1
Arm/Group | Enrolled, Received arTregs
Number analyzed (Participants) | 0

7. Secondary Outcome: Severity of Biopsy-Proven Acute Rejection (AR) and/or Clinical Rejection Events at Any Time After Alloantigen-Reactive Tregs (arTreg) Infusion
Description: Intensity of AR and/or clinical rejection events will be graded.
  Definitions:
  * AR: Diagnosed in accordance with Banff global assessment criteria
  * Clinical Rejection: Participants who are treated empirically based on investigator clinical suspicion in cases where a biopsy is indeterminate or in rare cases, where a biopsy cannot be performed.
Time Frame: From arTreg infusion through completion of study participation
Population: as for outcome 1
Arm/Group | Enrolled, Received arTregs
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Chronic Rejection Events at Any Time After Alloantigen-Reactive Tregs (arTreg) Infusion
Description: Diagnosed in accordance with Banff global assessment criteria.
Time Frame: From arTreg infusion through completion of study participation
Population: as for outcome 1
Arm/Group | Enrolled, Received arTregs
Number analyzed (Participants) | 0

9. Secondary Outcome: Proportion of Participants Who Successfully Discontinue Tacrolimus
Description: Proportion of participants who, per protocol:
  * fulfill eligibility for tacrolimus withdrawal,
  * subsequently achieve their last dose of tacrolimus,
  * remain tacrolimus-free for ≥12 weeks,
  * their liver function tests, ALT and GGT, are ≤50 U/L,
  * and their liver biopsy performed between 12 to 26 weeks status post the last dose of tacrolimus fulfills biopsy findings* for minimization of immunosuppression.
    * Biopsy findings: Liver histology will be assessed by central pathology. Biopsy findings for minimization of immunosuppression, per protocol. Reference: Demetris AJ, Bellamy C, Hubscher SG, et al. 2016 Comprehensive Update of the Banff Working Group on Liver Allograft Pathology: Introduction of Antibody-Mediated Rejection. Am J Transplant 2016.
Time Frame: Post-transplant through Completion of Study Participation
Population: as for outcome 1
Arm/Group | Enrolled, Received arTregs
Number analyzed (Participants) | 0

10. Secondary Outcome: Duration of Operational Tolerance
Description: Durability of operational tolerance defined as the time from achieving the primary endpoint to immunosuppression (IS) reinitiation or to the end of trial participation.
Time Frame: Post-transplant through Completion of Study Participation
Population: as for outcome 1
Arm/Group | Enrolled, Received arTregs
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 1.8 years
Description: Prior to study stage 2, only confirmed cases of COVID-19 were collected. All AEs were collected from the time of informed consent obtain during study stage 2 until the participant completes study participation or until 30 days after he/she prematurely withdraws (without withdrawing consent) or is withdrawn from the study.
Groups:
- Enrolled Transplant Recipient, Did Not Receive arTregs: These participants were consented and enrolled into the study, but did not receive arTregs.
Arm/Group | Enrolled Transplant Recipient, Did Not Receive arTregs | Enrolled Living Donor
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/30 | 0/12
Other Adverse Events (participants affected / at risk) | 3/30 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Transplant Recipient, Did Not Receive arTregs (N=30) | Enrolled Living Donor (N=12)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Transplant Recipient, Did Not Receive arTregs (N=30) | Enrolled Living Donor (N=12)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor in February 2023 prior to any participant receiving the investigational product, arTregs. The study's low enrollment would not allow for study completion within the necessary timeframe.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT03654040/Prot_SAP_000.pdf